CLINICAL TRIAL: NCT02137291
Title: IPg2 Study - Left-sided Lung Isolation: Comparison of Twodevices
Brief Title: IPg2 Study: Left-sided Lung Isolation
Acronym: IPg2
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean Bussières, Anesthesiologist, Full clinical professor, Laval University
Other Study IDs: IUCPQ-20952
Record Dates: First submitted 2013-09-19; First posted 2014-05-13 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Video-assisted Thoracoscopic Surgery (VATS); One-lung Ventilation
Keywords: Video-assisted thoracoscopic surgery (VATS); Lung isolation device; One-lung ventilation; Double lumen endotracheal tube; Bronchial blocker

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Left-sided double-lumen tube: Lung isolation with a left-sided double-lumen tube (BronchoCath, Mallinckrodt Medical, Cornamaddy, Athlone, Westmeath, Ireland)
- Modified right-sided double-lumen tube: Right-sided double-lumen tube modified in accordance with Bussières et al. in Can J Anesth 2007

SUMMARY:
Lung isolation is primordial in thoracic surgery. To achieve it, two techniques are used: the double lumen tube (DLT) and the bronchial blocker (BB). Left-sided DLT (L-DLT) is use by the majority of anesthesiologists for both left and right thoracic surgeries. Standard right-sided DLT (Rs-DLT) is rarely use since it is dif¬ficult to properly position it and that there is a risk of misalignment between the lateral orifice of the tube and the origin of the right upper lobe (RUL) bron¬chus. In 2007, the investigators have published results suggesting enlarging the Rs-DLT's lateral orifice. The modified R-DLT (Rm-DLT) was more frequently in an adequate position: 77% vs 37% of patients (p = 0.0121), and easier to reposition: 97% vs 74% of patients (p= 0.0109) in comparison to the standard R-DLT group. The data suggest the superiority of the Rm-DLT compared to Rs-DLT for optimal positioning to facilitate one-lung ventilation (OLV) during thoracic surgery. It is believed that DLT tend to provide quicker and better quality of lung collapse than BB. In 2013, investigators have demonstrated an equivalent quality of lung collapse (LC) between L-DLT and BB used with two apnea periods when initiating OLV. Complementary analysis showed a significative difference to obtain complete LC (CLC) between L-DLT for left thoracoscopy and L-DLT for right thoracoscopy and BB in right or left surgery. The investigator hypothesis is that, when using L-DLT for left video-assisted thoracoscopic surgery (VATS), LC of the isolated lung will be slower and of poorer quality compare to the use of the Rm-DLT. The primary objective is to compare the delay between pleural opening (PO) and CLC in left VATS when using three lung isolation devices: 1) L-DLT and 2) Rm-DLT. Secondary objectives are: 1) to evaluate quality of LC, 2) to evaluate the level of obstruction of the lumen of the left bronchus, 3) to evaluate the quality of OLV (PaO2) 4) To collect blind surgeon's opinion about de device used and 5) to measure the delay between OLV and PO for evaluating the role of absorption atelectasis in obtaining CLC. After obtaining IRB approval, the investigators propose a study of 40 patients undergoing an elective left VATS at IUCPQ involving one lung ventilation. They will have to be 21 years or more, to read, understand and sign an informed consent at their pre-operative evaluation. This study will be prospective, randomized, and blind to thoracic surgeons.

DETAILED DESCRIPTION:
Background:

Lung isolation is frequently used in thoracic surgery. The quality of the isolation is crucial, especially for video-assisted thoracoscopic surgery (VATS). Two techniques are principally used to obtain lung isolation: the double lumen tube (DLT) and the bronchial blocker (BB).

The left-sided DLT (L-DLT) is used by the majority of anesthesiologists, as much for left as for right thoracic surgeries. The standard right-sided DLT (Rs-DLT) is rarely used since positioning its lateral orifice with the origin of the right upper lobe (RUL) can be difficult.(1-4) In 2007, the investigators have published their results suggesting an enlargement of the lateral orifice of the Rs-DLT.(5) They have demonstrated that the modified right-sided double lumen tube (Rm-DLT) remained more frequently in optimal position than the Rs-DLT (77% vs. 37%, p=0.0121) and that it was also easier to reposition the tube after turning the patient in lateral decubitus (97% vs. 74%, p=0.0109).

More recently, investigators have demonstrated, with three dimensional reconstruction of computed tomography of 106 patients, that angulation between the RUL and the horizontal posterior plane varies from -26 to +58°, justifying the modification of the Rs-DLT proposed in 2007. (Unpublished data)

The use of BB for lung isolation is believed to provide a slower and a poorer quality of lung collapse (LC) than DLT. Over the years, the investigators have demonstrated an equivalent quality of lung collapse between the L-DLT and BB when two apnea periods are used at the beginning of one-lung ventilation (OLV). (Unpublished data) Further to complementary analysis, investigators have noted a significant difference in time to get complete lung collapse between left and right thoracic surgery when using the L-DLT. Time to obtain complete lung collapse (CLC) was not different when comparing BB and L-DLT in left thoracic surgery.

The hypothesis to explain these observations is that when the bronchial extremity of the L-DLT is inserted into the left main stem bronchus (LMSB), the LMSB and its relative superior position, associated to a progressive collapse of the left lung, could induce a dynamic obstruction of the distal extremity of the L-DLT lumen, and consequently slowing the lung collapse. Investigators have also regularly observed this type of obstruction during bronchoscopic examination when positioning the L-DLT.

In past studies comparing L-DLT to BB, time to get CLC was measured from the beginning of OLV. Nevertheless, the interval between this time point and the pleural opening (PO) is sometime difficult to control. Technical incidents can prolong this period and induce a bias. Furthermore, in the last investigator's protocol, the second period of apnea is done at pleural opening. For these reasons, the authors consider that the time to get CLC should be measured from the pleural opening since it is the crucial moment for the surgical team. Investigators are proposing to evaluate the PO-CLC interval as a primary objective.(6)

Hypothesis:

The hypothesis of the proposed study is that the use of the L-DLT will allow for a slower and a poorer quality of CLC compared to the ones obtained with the Rm-DLT in left VATS.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* elective left video-assisted thoracoscopy
* one lung ventilation

Exclusion Criteria:

* Anticipated difficult mask ventilation or intubation
* tracheal or high bronchial origin of the right upper lobe main bronchus
* severe COPD or asthma
* pleural disease
* previous left thoracic surgery
* chest radiotherapy
* chimiotherapy
* significant systemic co-morbidity
* active or chronic pulmonary infection
* fibrosis, other interstitial diseases
* endobronchial mass
* tracheostomy
* severe desaturation in the peroperative period
* any clinical situation precluding the use of an isolation device

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing an elective left VATS requiring OLV
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Time to obtain complete lung collapse | Peroperative
  Time to obtain complete lung collapse will be collected from the pleural opening up to complete lung collapse.

SECONDARY OUTCOMES:
Quality of lung collapse | Peroperative
  Quality of lung collapse from de beginning of one-lung ventilation to the end of surgery
Degree of obstruction of the right upper lobe bronchus lumen | Peroperative
  Degree of obstruction of the right upper lobe bronchus lumen from de beginning of one-lung ventilation to the end of surgery
Quality of one-lung ventilation | Peroperative
  Quality of one-lung ventilation from de beginning of one-lung ventilation to the end of surgery
Thoracic surgeon's guess about the device used | Peroperative
  Thoracic surgeon must guess which device was used by the anesthesiologist to isolate the lung 20 minutes after pleural opening. Choice: 1= L-DLT or 2= Rm-DLT
Time between the beginning of one-lung ventilation to pleural opening | Peroperative
  Time between the beginning of one-lung ventilation to pleural opening from de beginning of one-lung ventilation to the pleural opening

CONTACTS AND LOCATIONS:
Overall Officials: Jean S Bussières, MD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada

REFERENCES:
- [Background] Slinger P. The clinical use of right-sided double-lumen tubes. Can J Anaesth. 2010 Apr;57(4):293-300. doi: 10.1007/s12630-009-9262-z. No abstract available. English, French. PMID 20058114
- [Background] McKenna MJ, Wilson RS, Botelho RJ. Right upper lobe obstruction with right-sided double-lumen endobronchial tubes: a comparison of two tube types. J Cardiothorac Anesth. 1988 Dec;2(6):734-40. doi: 10.1016/0888-6296(88)90096-8. PMID 17171882
- [Background] Bussieres JS, Lacasse Y, Cote D, Beauvais M, St-Onge S, Lemieux J, Soucy J. Modified right-sided Broncho-Cath double lumen tube improves endobronchial positioning: a randomized study. Can J Anaesth. 2007 Apr;54(4):276-82. doi: 10.1007/BF03022772. PMID 17400979
- [Background] Ko R, McRae K, Darling G, Waddell TK, McGlade D, Cheung K, Katz J, Slinger P. The use of air in the inspired gas mixture during two-lung ventilation delays lung collapse during one-lung ventilation. Anesth Analg. 2009 Apr;108(4):1092-6. doi: 10.1213/ane.0b013e318195415f. PMID 19299766
- [Background] Brodsky JB, Lemmens HJ. Tracheal width and left double-lumen tube size: a formula to estimate left-bronchial width. J Clin Anesth. 2005 Jun;17(4):267-70. doi: 10.1016/j.jclinane.2004.07.008. PMID 15950850
- [Background] Fortier G, Cote D, Bergeron C, Bussieres JS. New landmarks improve the positioning of the left Broncho-Cath double-lumen tube-comparison with the classic technique. Can J Anaesth. 2001 Sep;48(8):790-4. doi: 10.1007/BF03016696. PMID 11546721